CLINICAL TRIAL: NCT03134898
Title: Longitudinal Study to Identify Predictive Factors of Post-thrombotic Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Ferran Barbe, Ferran Barbé, Hospitales Universitarios Virgen del Rocío
Other Study IDs: OSIRIS
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Hypertension; Pulmonary Thromboembolisms
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current data on the incidence of pulmonary hypertension (PH) are very variable, depending on the different studies designs. There are no data on the prognostic of PH in patients with asymptomatic pulmonary thromboembolisms (PT), neither paucisymptomatic PH, in which without a prospective follow-up would be underdiagnosed. We thought that the prognosis of both clinical forms (PT with or without symptoms) would be similar.

The objective of this study is know the real incidence of pulmonary hypertension (PH) post symptomatic and asymptomatic pulmonary thromboembolic (PT).

DETAILED DESCRIPTION:
Rationale

Pulmonary hypertension (PH) post pulmonary thromboembolisms is a serious and complex disease, is one major cause of pulmonary hypertension (1). It is the most feared late complication of pulmonary thromboembolism (PT) characterized by the organization of thrombotic material within the pulmonary arteries (2). Although a purely mechanical theory is too simplistic in view of the lack of correlation between the proportion of obliterated pulmonary arteries and the numbers of PH.

Acute, symptomatic, or asymptomatic PT may be the initial event, but disease progression would result from progressive vascular remodeling of small vessels. It is possible that unresolved pulmonary arterial thrombosis is a decisive factor for vascular endothelial cells to initiate their mesenchymal transition (3).

On the other hand, Pulmonary hypertension post pulmonary thromboembolisms is the only subclass of pulmonary hypertension that has a curative surgical treatment (4). The diagnosis of this situation should be detected as soon as possible to optimize the results of surgical and pharmacological treatment. Surgical indication should be established as early as possible to avoid progression (5).

Hypothesis

The current data on the incidence of PH are very variable, depending on the different studies designs. There are no data on the prognostic of PH in patients with asymptomatic PT, neither paucisymptomatic PH, in which without a prospective follow-up would be underdiagnosed. We thought that the prognosis of both clinical forms (PT with or without symptoms) would be similar. Also we thought and that there are forms of paucisymptomatic PH whose diagnosis and treatment would benefit from a prospective follow-up.

Objectives

Main objective

To know the incidence of pulmonary hypertension (PH) post symptomatic and asymptomatic pulmonary thromboembolic (PT).

The secondary objectives of the study are:

* To defined clinical subtypes of PT with a predictive value of diagnosis of PH in two years.
* To Measure biomarkers described that may be related to the diagnosis of PH or the disease progression.
* Use of genetic, proteomic, RNA transcription, cytometric and cellular and metabolic identification assays to aid in the search for new genetic factors and / or PH biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older and able to provide informed consent
* Diagnosis of pulmonary thromboembolisms confirmed by
* Computed Tomography Angiography (CTA) if there are a partial transluminal defect surrounded by contrast or a complete occlusion of pulmonary artery.
* Pulmonary ventilation/perfusion scan.- Patients with high risk based on PIOPED study criteria or in patients with deep venous thrombosis confirmed by echography and positron emission tomography (PET) scan not concluding.

Exclusion Criteria:

* Any contraindication to the performance of the pulmonary hypertension diagnostic tests
* Any circumstance, to investigator criteria, to impede the patient follow up
* Life expectancy lower than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diagnosis of incidental or symptomatic pulmonary thromboembolisms
Sampling Method: Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2013-11-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary hypertension | 2 years
  Diagnosis on pulmonary hypertension after pulmonary thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Remedios Otero Candelera, Study Chair — Hospital Universitario Virgen del Rocío IBIS
Locations (23):
- Spain (23):
  - Hospital M. de Badalona, Badalona, Barcelona
  - Hospital U. German Trias i Pujol, Badalona, Barcelona
  - Hospital G. de Cataluña, Sant Cugat del Vallès, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital U. Marqués de Valdecilla, Santander, Cantabria
  - Hospital Sierrallana, Torrelavega, Cantabria
  - Hospital de Cruces, Bilbao, Guipuzcua
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital U. Fundación Alcorcón, Alcorcón, Madrid
  - Hospital U. de Getafe, Getafe, Madrid
  - Hospital Virgen del Camino, Pamplona, Navarre
  - Hospital U. Central. de Asturias, Oviedo, Principality of Asturias
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Hospital de Araba, Alava
  - Hospital del Mar, Barcelona
  - Hospital U. de Girona Doctor Josep Trueta, Girona
  - Hospital U. Virgen de las Nieves, Granada
  - Hospital U. La Paz, Madrid
  - Hospital U. Ramón y Cajal, Madrid
  - Hospital San Juan de Dios, Seville
  - Hospital C. U. de Valladolid, Valladolid
  - Hospital C. U. Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tueller C, Stricker H, Soccal P, Tamm M, Aubert JD, Maggiorini M, Zwahlen M, Nicod L; Swiss Society for Pulmonary Hypertension. Epidemiology of pulmonary hypertension: new data from the Swiss registry. Swiss Med Wkly. 2008 Jun 28;138(25-26):379-84. doi: 10.4414/smw.2008.11915. PMID 18587690
- [Background] Lang IM. Chronic thromboembolic pulmonary hypertension--not so rare after all. N Engl J Med. 2004 May 27;350(22):2236-8. doi: 10.1056/NEJMp048088. No abstract available. PMID 15163772
- [Background] Humbert M. Pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension: pathophysiology. Eur Respir Rev. 2010 Mar;19(115):59-63. doi: 10.1183/09059180.00007309. PMID 20956167
- [Background] Condliffe R, Kiely DG, Gibbs JS, Corris PA, Peacock AJ, Jenkins DP, Hodgkins D, Goldsmith K, Hughes RJ, Sheares K, Tsui SS, Armstrong IJ, Torpy C, Crackett R, Carlin CM, Das C, Coghlan JG, Pepke-Zaba J. Improved outcomes in medically and surgically treated chronic thromboembolic pulmonary hypertension. Am J Respir Crit Care Med. 2008 May 15;177(10):1122-7. doi: 10.1164/rccm.200712-1841OC. Epub 2008 Feb 21. PMID 18292468
- [Background] Galie N, Kim NH. Pulmonary microvascular disease in chronic thromboembolic pulmonary hypertension. Proc Am Thorac Soc. 2006 Sep;3(7):571-6. doi: 10.1513/pats.200605-113LR. PMID 16963536
- [Derived] Otero R, Lobo JL, Lopez R, Fernandez C, Jimenez D, Muriel A, Alfonso M, Ballaz A, Nunez-Ares A, Rodriguez-Matute C, de Miguel-Diez J, Rodriguez-Chiaradia DA, Alcalde M, Elias T, Jara-Palomares L, Rivas A, Alonso A, Garcia-Ortega A, Sancho T, Morillo R, Garcia-Bragado F, Hernandez-Blasco L, Uresandi F, Madridano O, Aguero R, Monreal M; OSIRIS Investigators. Feasibility of a screening algorithm for chronic thromboembolic pulmonary hypertension: The OSIRIS study. Thromb Res. 2023 Aug;228:1-9. doi: 10.1016/j.thromres.2023.05.005. Epub 2023 May 19. PMID 37263121